CLINICAL TRIAL: NCT03989362
Title: Phase 2 Multicenter Trial of ICOS Agonist Monoclonal Antibody (mAb) Vopratelimab (JTX -2011) and a CTLA-4 Inhibitor in PD-1/PD-L1 Inhibitor Experienced Adult Subjects With Non-small Cell Lung Cancer or Urothelial Cancer
Brief Title: Vopratelimab and a CTLA-4 Inhibitor in PD-1/PD-L1 Inhibitor Experienced Subjects With NSCLC or Urothelial Cancer
Acronym: EMERGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jounce Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JTX-2011-201
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-04

CONDITIONS: Cancer
Keywords: ICOS; ICOS agonist monoclonal antibody; JTX-2011; Vopratelimab; Anti-CTLA-4; Ipilimumab; EMERGE; Immunotherapy; Immuno-Oncology; Cancer; Non-small Cell Lung Cancer; Urothelial Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LM1 (Experimental): Phase 2 study of vopratelimab by intravenous (IV) infusion administered in combination with ipilimumab by IV infusion in NSCLC
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- LT1 (Experimental): Phase 2 study of vopratelimab by IV infusion administered in combination with ipilimumab by IV infusion in NSCLC
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- UM1 (Experimental): Phase 2 study of vopratelimab by IV infusion administered in combination with ipilimumab by IV infusion in urothelial cancer
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- UT1 (Experimental): Phase 2 study of vopratelimab by IV infusion administered in combination with ipilimumab by IV infusion in urothelial cancer
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- LM2 (Experimental): Phase 2 study of vopratelimab by intravenous (IV) infusion in administered in sequence with ipilimumab by IV infusion in NSCLC
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- LT2 (Experimental): Phase 2 study of vopratelimab by intravenous (IV) infusion in administered in sequence with ipilimumab by IV infusion in NSCLC
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- UM2 (Experimental): Phase 2 study of vopratelimab by intravenous (IV) infusion in administered in sequence with ipilimumab by IV infusion in urothelial cancer
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab
- UT2 (Experimental): Phase 2 study of vopratelimab by intravenous (IV) infusion in administered in sequence with ipilimumab by IV infusion in urothelial cancer
  Interventions: Drug: Vopratelimab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Vopratelimab — Specified dose on specified days
  Other Names: JTX-2011
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy

SUMMARY:
JTX-2011-201 is a Phase 2, open label clinical study of vopratelimab (JTX-2011) and ipilimumab in adult subjects with non-small cell lung cancer (NSCLC) or urothelial cancer to evaluate safety and efficacy.

DETAILED DESCRIPTION:
Vopratelimab (JTX-2011) is an agonist monoclonal antibody that specifically binds to the Inducible CO-Stimulator of T cells (ICOS) to generate an anti-tumor immune response. This is a Phase 2, open label study to evaluate the safety and efficacy of vopratelimab in combination with ipilimumab in adult subjects with advanced and/or refractory non-small cell lung cancer and urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to participate and comply with all trial requirements and able to provide signed and dated informed consent prior to initiation of any trial procedures
2. Male or female ≥ 18 years of age
3. Locally advanced, inoperable or metastatic NSCLC or urothelial cancer, with evaluable or measurable disease, according to RECIST v1.1, with at least one measurable lesion
4. Prior treatment with a PD-1/PD -L1 inhibitor for at least 3 months
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Predicted life expectancy ≥ 3 months
7. Have laboratory values in accordance with the study protocol
8. If medical history of the following, case should be reviewed with the Medical Monitor: prior biliary tract disorders (as based on Hepatobiliary system organ class high level terms of obstructive bile duct disorders, hepatic vascular disorders, structural and other bile duct disorders) or portal hypertension and/or hepatic vascular disorders
9. Women of child-bearing potential (WOCBP): negative serum pregnancy test within 72 hours prior to planned C1D1 and a negative urine pregnancy test on C1D1 and any subsequent study drug administration day
10. WOCBP and males whose partners are WOCBP must agree to use a highly effective method of birth control throughout their participation and for 5 months following the last study drug administration. Highly effective methods of birth control are defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1 percent per year) when used consistently and correctly. For subjects using a hormonal contraceptive method, information regarding the product under evaluation and its potential effect on the contraceptive should be addressed.

Exclusion Criteria:

1. Concurrent anticancer treatment (either approved or investigational, excluding radiation therapy)
2. Prior anticancer therapies within the timeframes specified below, or ongoing toxicity from prior therapy > Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Exceptions include > Grade 1 toxicities that, in the opinion of the Investigator, should not exclude the subject (e.g., alopecia) and are approved by the Medical Monitor:

   1. Biologic therapy, including immunotherapy, within 21 days prior to C1D1
   2. Chemotherapy within 21 days (42 days for mitomycin or nitrosoureas) prior to C1D1
   3. Anti-CTLA-4 or anti-ICOS therapy at any time
   4. Chimeric antigen receptor T-cell therapy at any time
   5. Organ transplantation, including allogeneic or autologous stem-cell transplantation, at any time
3. Major surgery (excluding minor procedures, e.g., placement of vascular access, biopsy, etc.) within 4 weeks prior to C1D1
4. Live vaccines within 30 days prior to C1D1 (inactivated vaccines are allowed; seasonal vaccines should be up to date prior to C1D1)
5. History of immune-related adverse events (irAEs) leading to treatment discontinuation. Subjects who discontinued prior immunotherapies for irAEs that are well controlled with appropriate treatment may be enrolled if approved by the Medical Monitor
6. Any active disease, including primary or acquired immunodeficiency, requiring systemic immunosuppressive therapy equivalent to ≥10 mg prednisone per day within 7 days prior to C1D1. Exception: inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease as well as a one-time dose of immunosuppressive agents used prophylactically for contrast allergies
7. Known severe intolerance to or life-threatening hypersensitivity reactions to humanized monoclonal antibodies or intravenous immunoglobulin preparations; history of anaphylaxis; or known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
8. Brain metastases, leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation
9. Prior whole brain radiation
10. Concurrent second malignancy at other sites that requires treatment or, in the judgment of the Investigator, may require treatment within the next year. Concurrent malignancies that do not require treatment and are clinically stable are allowed. Prior malignancies are allowed as long as the subject is not receiving specific treatment other than hormonal therapy and, in the judgment of the Investigator, is unlikely to have a recurrence
11. Active and clinically relevant bacterial, fungal, or viral infection, including known Hepatitis A, B, or C or human immunodeficiency virus (HIV) (testing not required)
12. Women who are pregnant or breastfeeding
13. History of symptomatic cardiac disease that is unresponsive to surgical or medical management
14. Any medical or social condition that, in the opinion of the Investigator, might place a subject at increased risk, affect compliance, or confound safety or other clinical trial data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
% subjects with overall response (OR) | 34 months

SECONDARY OUTCOMES:
% subjects with adverse events (AEs) | 34 months
% subjects with serious adverse events (SAEs) | 34 months
% subjects with clinically significant change from baseline in clinical laboratory tests | 34 months
% subjects with anti-drug antibodies (ADA) to treatment | 34 months
% of subjects with neutralizing antibodies (NAb) to treatment | 34 months
% of subjects with clinically significant changes in electrocardiogram (ECG) measurements | 34 months
Percent change in target lesions from baseline | 34 months
Apparent volume of distribution during specific time points | 34 months
Median duration of response (DOR) | 34 months
Disease control rate (DCR) | 34 months
Landmark progression free survival (PFS) | 34 months
Median PFS | 34 months
Median overall survival (OS) | 34 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Hooper, MD, Study Director — Jounce Therapeutics, Inc.
Locations (21):
- United States (18):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - University of Southern California Medical Center, Los Angeles, California
  - Christiana Care Health Services, Newark, Delaware
  - Florida Cancer Specialists Sarasota Cattlemen, Sarasota, Florida
  - University of Maryland - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - Weill Cornell Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - Southeastern Medical Oncology Center, Clinton, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of The Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (3):
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - The Research Institute of the McGill University Health, Montreal, Quebec
  - University Institute of Cardiology and Respirology of Quebec, Québec

IPD SHARING:
Plan to Share IPD: No